CLINICAL TRIAL: NCT01433757
Title: A Pilot, Randomized, Double-Blind, Placebo-Controlled Phase I Study to Determine the Safety and Efficacy of Ampicillin in Treating Primary Dystonia Symptoms
Brief Title: Ampicillin for DYT-1 Dystonia Motor Symptoms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Tyler's Hope for a Dystonia Cure, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 301-2011
Record Dates: First submitted 2011-08-05; First posted 2011-09-14 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: DYT-1; Dystonia
Keywords: dystonia; DYT-1; AMPICILLIN
MeSH Terms: conditions — Dystonia | interventions — Ampicillin; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ampicillin (Active Comparator): Patients who are randomly selected to receive the active drug will receive Ampicillin (2mg daily for adults and 1 mg daily for children).
  Interventions: Drug: Ampicillin
- Placebo (Placebo Comparator): Patients who are randomly selected to receive the placebo will be given a sugar pill that resembles the active drug.
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Ampicillin — Ampicillin will be given in capsule form. Dosage will be 2 mg daily for adults and 1 mg daily for children. One capsule will be taken each day for 28 consecutive days. After the first 28 days, there will be a 7 day 'washout' period during which no capsules are taken. Following the 'washout' period, another 28-day supply of Ampicillin will be given to the patient, to be taken in the same manner as described above.
  Arms: Ampicillin
Drug: Sugar pill — The sugar pill will be given in capsule form. Dosage will be 2 mg daily for adults and 1 mg daily for children. One capsule will be taken each day for 28 consecutive days. After the first 28 days, there will be a 7 day 'washout' period during which no capsules are taken. Following the 'washout' period, another 28-day supply of the sugar pill will be given to the patient, to be taken in the same manner as described above.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate if the antibiotic Ampicillin is safe and tolerated in patients that have generalized dystonia caused by the DYT-1 gene mutation, as compared to patients treated with a placebo. A placebo is a pill that looks and tastes the same as the real drug, but without the active ingredient. The second objective of this study is to determine if dystonia symptoms improve while on the study drug.

DETAILED DESCRIPTION:
This is a double-blinded and randomized drug study: neither the patient nor the investigator know if patients are taking study drug (Ampicillin) or placebo.

Three study visits will include neurological exams, review of medical history, genetic test results and video-taped BFM-DRS motor scales. Patients will receive medication during baseline visit, consisting of either Ampicillin drug or placebo, which will be consumed twice daily for 28 days. Following a washout period (no drugs) of 7 days, patient will return to clinic for second study visit and receive second set of medication (placebo -vs- Ampicillin). Medication will be consumed twice daily for 28 days, with patient returning to clinic after a washout period of 7 days for final study visit in clinic.

ELIGIBILITY:
Inclusion Criteria:

* DYT-1 dystonia, confirmed by genetic testing
* Between ages of 7 and 80 years
* BFM-DRS score greater than 6

Exclusion Criteria:

* Negative DYT-1 dystonia gene test
* Allergy to penicillins or cephalosporins
* Concurrent bacterial, viral or fungal infection at time of enrollment
* Pregnancy
* Inability to follow study protocol
* Lactose intolerance (placebo contains lactose powder)

Ages: 7 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-09; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of Ampicillin in treating DYT-1 dystonia | 70 days
  The primary objective of this study is to evaluate the safety and tolerability of treating DYT-1 dystonia with the use of ampicillin as compared to placebo.

SECONDARY OUTCOMES:
Burke-Fahn Marsden Dystonia Rating Scale (BFM-DRS) | 70 days
  We will determine if there is a reduction in Burke-Fahn Marsden Dystonia Rating Scale motor scores at the end of the study period and compare with the placebo treated group.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Malaty, M.D., Principal Investigator — University of Florida
Locations (1):
- UF Center for Movement Disorders and Neurorestoration, Gainesville, Florida, United States